CLINICAL TRIAL: NCT02592083
Title: PREDIX Luminal A - Neoadjuvant Response-guided Treatment of Slowly Proliferating Hormone Receptor Positive Tumors. Part of a Platform of Translational Phase II Trials Based on Molecular Subtypes
Brief Title: Neoadjuvant Response-guided Treatment of Slowly Proliferating Hormone Receptor Positive Tumors
Acronym: PREDIX LumA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Hatschek (Other)
Responsible Party: Sponsor-Investigator, Thomas Hatschek, Sen. Consultant, MD, PhD, Assoc. professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDIX LumA
Record Dates: First submitted 2015-10-26; First posted 2015-10-30 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Early-Stage Breast Carcinoma; Hormone Receptor Positive Tumor
Keywords: Neoadjuvant Therapy; Cyclin-Dependent Kinase Inhibitor p16
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Aromatase Inhibitors; Goserelin; Letrozole; Anastrozole; exemestane; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A: Endocrine treatment (Active Comparator): Pre- or perimenopausal women are treated with tamoxifen, alternatively with an LHRH analogue in combination with an aromatase inhibitor (only women); postmenopausal women receive an aromatase inhibitor. The preoperative treatment is continued for further 12 weeks, provided that re-evaluation after 6 weeks, week 10 of the preoperative treatment, does not indicate progression. Upon progression (PD), individualized management, preferentially surgery, is the primary option
  Interventions: Drug: Tamoxifen or Aromatase Inhibitor or Aromatase Inhibitor + goserelin
- B: Endocrine treatment + palbociclib (Experimental): Patients receive the same endocrine treatment as in arm A together with palbociclib 125 mg orally days 1-21, followed by a 7-days rest period. The combined treatment is continued for further 12 weeks, provided that re-evaluation after 6 weeks, week 10 of the preoperative treatment, does not indicate progression. Upon progression (PD), individualized management, preferentially surgery, is the primary option
  Interventions: Drug: Tamoxifen or Aromatase Inhibitor or Aromatase Inhibitor + goserelin; Drug: Palbociclib
- C: Endocrine treatment + palbociclib (Experimental): Patients receive the same endocrine treatment as in arm A together with palbociclib 125 mg orally days 1-21, followed by a 7-days rest period. The combined treatment is continued for further 12 weeks, if re-evaluation after 6 weeks, week 10 of the preoperative treatment, does not indicate progression. Upon progression (PD), individualized management, preferentially surgery, is the primary option
  Interventions: Drug: Tamoxifen or Aromatase Inhibitor or Aromatase Inhibitor + goserelin; Drug: Palbociclib

INTERVENTIONS:
Drug: Tamoxifen or Aromatase Inhibitor or Aromatase Inhibitor + goserelin
  Other Names: Tamoxifen; Letrozol or Anastrozol or Exemestane; Zoladex
Drug: Palbociclib
  Other Names: Ibrance
  Arms: B: Endocrine treatment + palbociclib; C: Endocrine treatment + palbociclib

SUMMARY:
The purpose of this neoadjuvant trial is to evaluate efficacy and toxicity of the cdk 4/6 inhibitor palbociclib when added to standard endocrine treatment. Initially, patients receive endocrine treatment for 4 weeks. In case of decrease of proliferation (Ki67) patients are then randomized between either continuous endocrine therapy (arm A) or the same treatment with addition of palbociclib (arm B). Patients with no change of proliferation are allocated to endocrine treatment + palbociclib without randomization (arm C). During the 12-weekly treatment period, clinical and radiological evaluations are performed repeatedly. Switch between the treatment arms A and B is allowed in case of lack of response or due to toxicity. A translational subprotocol is a mandatory part of the study protocol, except for use of PET-CT evaluations.

DETAILED DESCRIPTION:
Pre- or perimenopausal women are treated with tamoxifen, alternatively with an LHRH analogue in combination with an aromatase inhibitor (only women). Postmenopausal women receive an aromatase inhibitor.This treatment is given for 4 weeks. In cases with uncertain menopausal status (previous hysterectomy and equivocal gonadotropins), postmenopause age limit is defined as 55 years or older.

Ki67 is determined by FNA or core biopsy before start and after 2 weeks of treatment. After the initial 4-week period, patients with signs of response in terms of decrease of Ki67 by ≥20% are randomized to endocrine treatment either alone or in combination with the cdk 4/6 inhibitor palbociclib (arm A and B). Patients with tumors with stable disease, defined as <20% decrease or increase of Ki67 and without radiological indication of tumor progression at the 4-week evaluation are offered continuous endocrine treatment with the addition of palbociclib (arm C).

Dose regimen after 4 weeks of endocrine pretreatment:

Arm A: Pre- or perimenopausal women are treated with tamoxifen, alternatively with an LHRH analogue in combination with an aromatase inhibitor (only women). Postmenopausal women receive an aromatase inhibitor. The preoperative treatment is continued for further 12 weeks, provided that re-evaluation after 6 and 10 weeks of the preoperative treatment does not indicate progression. Upon progression (PD), individualized management, preferentially surgery, is the primary option.

Arm B: Patients receive the same endocrine treatment as in arm A together with palbociclib 125 mg orally days 1-21, followed by a 7-days rest period. The combined treatment is continued for further 12 weeks, if re-evaluation after 6 weeks, week 10 of the preoperative treatment, does not indicate progression. Upon progression (PD), individualized management, preferentially surgery, is the primary option.

Arm C: Treatment according to the schedule as described for arm B.

Postoperative chemotherapy is recommended to patients with either residual lymph node metastases >2mm (macro metastases) or primary tumor size >30mm in combination with Ki67>15%. Adjuvant endocrine treatment and radiotherapy is offered according to standard guidelines. Structured follow-up visits yearly for five years include reporting of persistent treatment-related toxicity, HRQoL, recurrence and death.

All patients are recommended adjuvant endocrine treatment for at least 5 years.

The trial contains also a translational subprotocol:

1. PET-CT using FDG, confined to the chest, is performed before start of the first treatment period and after 10 weeks, i.e. 6 weeks after treatment allocation (functional imaging, optional).
2. Core biopsies from the tumor are collected before start of the first treatment period and after 10 weeks, i.e. 6 weeks after treatment allocation. Further tissue samples are collected from the surgical specimen.
3. Blood samples are collected repeatedly during the ongoing treatment and yearly follow-up.
4. FNAs from metastases in case of recurrence during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Female patients with non-lobular breast cancer confirmed by histology
3. Tumor and blood samples available. Luminal A type confirmed by immunohistochemistry with ER and PR positive ≥50% and the proliferation marker Ki 67 <20% and not HER2 amplified
4. Age older than 40 years
5. Primary breast cancer >20mm without lymph node metastases
6. Adequate bone marrow, renal, hepatic and cardiac functions and no other uncontrolled medical or psychiatric disorders
7. LVEF >50%
8. ECOG performance status 0-1

Exclusion Criteria:

1. Metastases, including node metastases in the ipsilateral and/or contralateral thoracic region or in the mediastinum
2. Other malignancy diagnosed within the last five years, except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix
3. Age ≤40 years
4. Lobular carcinoma
5. Patients in child-bearing age without adequate contraception
6. Pregnancy or lactation
7. Severe medical or psychiatric disorders where the study treatment or study procedures carry increased risk of deterioration of health status

Min Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2019-02 (Actual); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Clinical and Radiological Response | After 16 weeks of preoperative treatment
  Clinical evaluations by use of calliper, radiological evaluations with mammography and ultrasound after 4, 10 and 16 weeks, PET-CT after 10 weeks of treatment, compared with baseline measurements

SECONDARY OUTCOMES:
Pathological Evaluation of Tumor Response | From date of surgery up to 4 weeks
  Pathological signs of response, i.e. fibrosis, necrosis aso.
Disease-free Survival | From date of surgery until 60 months past surgery
  Disease-free survival includes all events related to breast cancer, and death from any cause during the follow-up period
Breast Cancer-specific Survival | From date of surgery until 60 months past surgery
  Breast cancer-specific survival includes all events related to breast cancer and death caused by breast cancer during the follow-up period
Overall Survival | From date of surgery until 60 months past surgery
  Overall survival relates to death from any cause during the follow-up period
Incidence of treatment-emergent adverse events [Safety and Tolerability] | From start of treatment until 28 days after termination of treatment. Delayed toxicity is reported until 60 months follow-up
  Safety will be assessed using NCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE) for reporting laboratory and non-laboratory toxicities.
Health-related Quality of Life | From start of study treatment until termination, and then annually during the 60 months of postoperative follow-up period
Biological characteristics of tumors exposed to targeted treatment of early breast cancer | Before start and during treatment, at surgery, and then annually during the 60 months of postoperative follow-up period
  Includes core biopsies and blood samples before start and after 10 weeks of treatment, collection of tumor samples from the surgical specimen at the date of operation, blood samples in connection with annual follow-up visits and FNA and blood samples in case of recurrence. Time frame for collection of biological samples from start of preoperative treatment until 60 months of follow-up post surgery. Planned analyses cover genomics (New Generation Sequencing) and proteomics
Immunohistochemical characteristics | Before start, during treatment and at the date of operation
  Includes core biopsies before start and after 10 weeks of treatment, and collection of tumor samples from the surgical specimen at surgery
Thymidine kinase (TK1) activity during study treatment | Before start and until termination of the preoperative treatment
  Includes repeated blood samples before start and after 4, 10 and 16 weeks of treatment
Drug metabolism during study treatment | Four and ten weeks after start of the preoperative treatment
  Includes repeated blood samples after 4 and 10 weeks of treatment with the aim to compare intra- and inter-patient metabolism of endocrine treatment in relation to response

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hatschek, Assoc. Prof., Study Chair — Breast-sarcoma Unit, Dept. of Oncology, Karolinska University Hospital; Jonas Bergh, Professor, Study Director — Dept. of Oncology-Pathology, Karolinska Institutet
Locations (1):
- Department of Oncology, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No